CLINICAL TRIAL: NCT03258489
Title: Effects of Transcutaneous Nervous Electric Stimulation (TENS) and Interferential Electrical Stimulation (IES) on the Autonomous Balance of Normotens Volunteers and Hypertensive Patients
Brief Title: Effects of TENS and IES on the Autonomous Balance of Normotens Volunteers and Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Luis Ulisses Signori, Principal Investigador, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFSM
Record Dates: First submitted 2017-07-26; First posted 2017-08-23 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers; Hypertension, Essential
MeSH Terms: conditions — Essential Hypertension | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous nervous electric stimulation (TENS) (Active Comparator): Autonomic balance, blood pressure, and blood collection (catecholamines) will be evaluated before and after TENS. The autonomic balance will be evaluated by heart rate variability (HRV), systemic arterial pressure (SBP) will be evaluated by an Ambulatory Blood Pressure Monitor (ABPM) and catecholamines of kits.
  Interventions: Device: Transcutaneous nervous electric stimulation (TENS)
- Interferential electrical stimulation (IES) (Active Comparator): Autonomic balance, blood pressure, and blood collection (catecholamines) will be evaluated before and after Interferential electrical stimulation (IES). The autonomic balance will be evaluated by heart rate variability (HRV), systemic arterial pressure (SBP) will be evaluated by an Ambulatory Blood Pressure Monitor (ABPM) and catecholamines of kits.
  Interventions: Device: Interferential electrical stimulation (IES)
- TENS and IES Placebo (Placebo Comparator): Autonomic balance, blood pressure, and blood collection (catecholamines) will be evaluated before and after of the TENS and IES placebo. The autonomic balance will be evaluated by heart rate variability (HRV), systemic arterial pressure (SBP) will be evaluated by an Ambulatory Blood Pressure Monitor (ABPM) and catecholamines of kits.
  Interventions: Device: TENS and IES Placebo

INTERVENTIONS:
Device: Transcutaneous nervous electric stimulation (TENS) — TENS (Frequency 10 Hz or 100Hz /duration 200μs, Endophasys nms 0501® model, KLD Biosystems, Amparo, SP, Brazil) will be applied with intensity between 1 to 60 mA and the current will be adjusted every 5 minutes at the sensory threshold level muscle contraction or according to the tolerance to the stimulus informed by the volunteers. TENS will be applied in bilateral paravertebral region of C7 to T4 or long the brachial plexus and sciatic plexus.
  Arms: Transcutaneous nervous electric stimulation (TENS)
Device: Interferential electrical stimulation (IES) — The IES (Endophasys nms 0501®, KLD Biosystems, Amparo, SP, Brazil) will be applied in continuous mode with biphasic pulses. Bipolar electrodes with slope of 1/5/1. The rest of the parameters will be set to 4000 Hz, AMF of 100 Hz and the AMF variation of 25 Hz. The effect of the current will be adjusted by the intensity, it should produce paresthesia stimuli, without pain and below the motor threshold. Adhesive electrodes (MultiStick®, Axelgaard Manufacturing CO, Ltd, Fallbrook, CA, USA) will be housed in the paravertebral region, between C7 (Channel 1) and T4 (Channel 2). (SANTOS et al., 2013)
  Arms: Interferential electrical stimulation (IES)
Device: TENS and IES Placebo — Same protocol without electrical output.
  Arms: TENS and IES Placebo

SUMMARY:
Hypertension is considered a serious public health problem. The imbalance in autonomic nervous system (ANS) activity is one of the main triggers in the development and maintenance of hypertension. The non-pharmacological management of this disease is an important resource, especially in refractory hypertensive patients or in hypertensive crises, where the pharmacological treatment does not present an efficient response. It is known that transcutaneous electrical nerve stimulation (TENS) is capable of modifying the autonomic balance, however, the effects of Interferential electrical stimulation (IES) on this system in normotensive and hypertensive volunteers are not yet known. These electrotherapeutic resources may be a non-pharmacological tool supporting the management of hypertension. The objective of this research is to study the effects of different TENS and IC parameters on cardiovascular variables of normotensive volunteers and hypertensive patients.

DETAILED DESCRIPTION:
Each volunteer will perform three assessments with a one-week interval. Each assessment will include assessment of autonomic balance, blood pressure, and blood collection (catecholamines). Interventions (placebo, low frequency TENS and IES) will be randomized. Volunteers will be accommodated in the supine position. With properly sanitized skin (70% alcohol) and self-adhesive electrodes (5x5 area) will be positioned in the cervical paravertebral region. All participants will be submitted to a placebo TENS session, a low frequency TENS session (TENS, 10 Hz/200μs) and an IES session (STEIN et al., 2012). The sessions will take place in the morning in a 12-hour fast, lasting 30 minutes, in an air-conditioned place (23ºC).

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Normal blood pressure (PAS <130 mmHg; PAD <85 mmHg) or Previous Hypertension diagnosis, systolic blood pressure (SBP) > 140 mm Hg and/or diastolic blood pressure (DBP) >90 mm Hg and clinical stability with no change in medications for at least 2 months preceding the study;
* The subjects that joined the study will be alphabetized volunteers;
* Age between 20 and 65 years old;
* With no symptoms of skeletal muscle disorders;
* No previous performing cardiovascular surgery;
* No previous diagnose of rheumatic, neurological, oncological, immune or hematologic diseases;
* Without evidence of psychiatric diseases and/or cognitive déficit;
* Non-Smoker;
* Volunteers with a body mass index (BMI: kg/m2) greater than 35 will not be included in the study

Exclusion Criteria:

* On the day of the assessments who have consumed of the alcoholic drink, caffeine and citrus juice and who have performed intense physical activities 48 before the examination

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Systemic arterial pressure (mmHg) | SBP will be evaluated 1 hours after the interventions
  Systemic arterial pressure (SBP) will be evaluated by an Ambulatory Blood Pressure Monitor (ABPM) (NOBRE et al., 2011). Micromed and version 5.0.1.52 equipment will be used. Blood pressure monitoring using ABPM will be performed every 10 min throughout the experiment, which has an estimated time of two hours.

SECONDARY OUTCOMES:
Blood collection - catecholamines (pg/mL) | Blood collection (catecholamines) will be evaluated 1 hours after the interventions
  Plasma levels of catecholamines (dopamine, epinephrine and norepinephrine) will be evaluated before and after HPLC (High Performance Liquid Chromatography) interventions. Blood with heparin will be homogenized and immediately transferred to a special tube containing 120 μL of EGTA/GSH (reduced glutathione) solution. After being centrifuged and the plasma transferred to a plastic tube, it is placed in a freezer (-80ºC).
Heart Rate Variability (n.u.) | HRV will be evaluated 1 hours after the interventions
  The autonomic balance evaluate by heart rate variability (HRV) and the heart rate signal will be purchased through a pulse frequency meter mark Polar model 810i (GAMELIN et al., 2006). The acquisition of ECG signal (sample rate-1 kHz) of the time series of RR will be purchased in continuous intervals (10 min). Data Will be transferred to a computer and RR intervals. They will be processed to calculate HRV parameter using the HRV analysis software KUBIOS. HRV will be analyzed in the time and frequency domain, using the area of greatest stability in RR intervals corresponding to 5 min of recordings (containing at least 256 consecutive beats) during controlled breathing. Volunteers Will remain in a supine position at rest for 10 min and afterwards, data will be collected with controlled breathing (12 breaths per minute; I/E:2/3) (STEIN et al., 2011). Values expressed in Total Power (ms2) and normalization unit (n.u.) (GAMELIN et al., 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Ulisses Signori, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gamelin FX, Berthoin S, Bosquet L. Validity of the polar S810 heart rate monitor to measure R-R intervals at rest. Med Sci Sports Exerc. 2006 May;38(5):887-93. doi: 10.1249/01.mss.0000218135.79476.9c. PMID 16672842
- [Result] Santos FV, Chiappa GR, Vieira PJ, Umpierre D, Ribeiro JP, Cipriano G Jr. Interferential electrical stimulation improves peripheral vasodilatation in healthy individuals. Braz J Phys Ther. 2013 May-Jun;17(3):281-8. doi: 10.1590/s1413-35552012005000092. PMID 23966145
- [Result] Sociedade Brasileira de Cardiologia (SBC); Sociedade Brasileira de Hipertensao (SBH); Sociedade Brasileira de Nefrologia (SBN). [V Guidelines for ambulatory blood pressure monitoring (ABPM) and III Guidelines for home blood pressure monitoring (HBPM)]. Arq Bras Cardiol. 2011 Sep;97(3 Suppl 3):1-24. No abstract available. Portuguese. PMID 22262107
- [Result] Stein C, Dal Lago P, Ferreira JB, Casali KR, Plentz RD. Transcutaneous electrical nerve stimulation at different frequencies on heart rate variability in healthy subjects. Auton Neurosci. 2011 Dec 7;165(2):205-8. doi: 10.1016/j.autneu.2011.07.003. Epub 2011 Aug 9. PMID 21827970
- [Result] Stein C, Mea Plentz RD. The effect of transcutaneous electrical nerve stimulation on blood pressure. Blood Press. 2013 Jun;22(3):188-9. doi: 10.3109/08037051.2012.722271. Epub 2012 Sep 25. No abstract available. PMID 23004921